CLINICAL TRIAL: NCT04151602
Title: Transmission of Tuberculosis Among Illicit Drug Use Linkages
Acronym: TOTAL
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: University of Stellenbosch (Other); Desmond Tutu HIV Foundation (Other); Boston University (Other); Medical Research Council, South Africa (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-38910; 1R01AI147316-01 (NIH)
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis; Illicit Drug Use
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum, exhaled bio-aerosols
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PWUD with active TB: People who use smoked illicit drugs (methamphetamine and/or methaqualone (mandrax)) with active TB disease
  Interventions: Behavioral: Smoked illicit drug use
- PWUD with no active TB: People who use smoked illicit drugs (methamphetamine and/or methaqualone (mandrax)) with no active TB disease
  Interventions: Behavioral: Smoked illicit drug use
- non-PWUD with active TB: People who do not use meth/mandrax who have active TB disease

INTERVENTIONS:
Behavioral: Smoked illicit drug use — The exposure of interest is current smoked illicit drug use, particularly methamphetamine and/or methaqualones
  Groups: PWUD with active TB; PWUD with no active TB

SUMMARY:
Tuberculosis (TB) is the leading infectious disease killer globally and leading cause of death in persons with HIV. The most effective way to reduce TB incidence and mortality is to interrupt transmission. This requires finding and treating individuals with TB disease early, including those with subclinical disease. Molecular epidemiologic studies and mathematical models have shown that the primary approach to case finding-household contact tracing-identifies only 8-19% of transmissions in high TB and TB/HIV burden settings. Thus there is a clear need to identify new groups and settings where TB transmission occurs. Spatial clustering of individuals with higher rates of progression from infection to disease, such as those with HIV and malnourishment, can also form transmission hotspots. Illicit drug (i.e., methamphetamines, crack/cocaine, opiates) users have higher TB infection prevalence and disease incidence compared to non-users, likely due to significant within-group transmission and/or clustered vulnerability. Increased transmission among people who use illicit drugs (PWUD) could result from creation of more efficient TB transmitters, increased close contact among transmitters, increased rates of primary progression from infection to disease among contacts, or a combination. Interrogation of illicit drug user networks for TB transmission, therefore, holds great potential as a target for early case identification and linkage to treatment, with potential benefit for halting transmission to the broader population.

DETAILED DESCRIPTION:
A cross-sectional, observational study design using respondent driven sampling (RDS) will be used for this research study.

In Aim 1, individuals will be recruited who currently use meth and/or Mandrax to assess TB exposure, incipient TB prevalence, and TB disease prevalence in the network. RDS will be used to seek out 750 meth/Mandrax users. Initial seeds (N=4) will be individuals from the investigator's current R01, the Tuberculosis treatment outcomes and alcohol use study (TRUST) cohort who have had active pulmonary TB disease in the prior 1-2 years and report current meth/Mandrax use.

For Aim 2, individuals from Aim 1 identified to have possible TB disease will be screened and enrolled to estimate the proportion that reflect recent transmission via genotyping and social epidemiologic links.

In Aim 3, the investigators will examine physiologic factors that may make PWUD more efficient TB transmitters. 50 PWUD participants from Aim 2 will be recruited who have active, untreated pulmonary TB and 50 individuals with active, untreated pulmonary TB who do not use meth/Mandrax, matched on age and gender will be recruited

ELIGIBILITY:
Participants must be/have the following general inclusion criteria:

1. at least 15 years old
2. resident of the study community
3. intact mental status at enrollment (i.e., no acute intoxication)
4. provide written, informed consent to participate in the study if ≥18 years or written assent and parental consent if <18 years.
5. agree to comply with all study requirements, including provision of contact information and study appointments attendance

And for Aim 1:

1. self-reported meth or Mandrax use in the past month
2. urine drug screen positive for meth and/or Mandrax
3. all participants other than the seeds must also have evidence that they have been recruited by a peer (the coupon)

For Aim 2 participants must meet all general inclusion criteria and the inclusion criteria from Aim 1 (meth/Mandrax use) and:

(1) Have evidence of active TB disease on Xpert Ultra from their Aim 1 visit testing or report a recent TB diagnosis (within the past month)

For Aim 3 Arm 1 participants must meet all general inclusion criteria and the criteria under Aim 1 and Aim 2 (active illicit drug use and active TB)

And exclusion criteria:

1. No current pregnancy by urine pregnancy test
2. Not yet started on TB medication

For Aim 3 Arm 2 patients must meet all general inclusion criteria and the following inclusion criteria:

1. Attend the Worcester Community Day Clinic, the Empilisweni Clinic, or any other clinic and live in the general Worcester area
2. Have newly diagnosed TB

And exclusion criteria:

1. No self-reported drug use or evidence of drug use by urine test
2. No current pregnancy by urine pregnancy test
3. Not yet started TB medication

General exclusion criteria under all aims and arms of the study include:

1. Current drug or alcohol intoxication
2. Mental incapacitation to providing informed consent
3. Not currently or previously enrolled in any prophylactic TB therapy studies

Participants may also be excluded from the study under discretion of the Principal Investigator if the PI believes participation in the study may prove harmful to the participant or the research staff.

Participants will be enrolled from the main cohort (n=750) (Aim 1) into the additional cohorts under Aims 2 and Aim 3 Arm 1. Aim 3 Arm 2 will be recruited external to the main cohort (Aim 1)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 750 PWUD in the Western Cape, South Africa will be enrolled into Aim 1. An anticipated 45-75 will have active TB disease and enrolled into Aim 2 and Aim 3 Arm 1 of the study.
  50 people who do not smoke illicit drugs with active TB disease will be enrolled into Aim 3 Arm 2.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
TB disease prevalence | At baseline
  Percentage of persons with TB disease based on results from Xpert Ultra and sputum culture
Incipient TB prevalence | At baseline
  Percentage of persons with incipient TB based on host RNA signature
Proportion of active TB cases resulting from recent transmission within this network of PWUD | At baseline
  Proportion of linked TB cases based on whole genome sequencing of the mycobacterium tuberculosis (Mtb) isolate and overlaying social epidemiological ties
Quantity of aerosolized Mtb in exhaled breath: amount of aerosolized Mtb exhaled in one hour | One hour
  The amount of aerosolized Mtb exhaled in one hour in a specialized bio-aerosol capturing booth

CONTACTS AND LOCATIONS:
Overall Officials: Karen Jacobson, MD MPH, Principal Investigator — Boston Medical Center/ BUMC
Locations (1):
- Privately Rented Facility, Worcester, South Africa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04151602/ICF_000.pdf